CLINICAL TRIAL: NCT02888106
Title: A Multicenter, Open-label, Randomised, Comparative, Parallel-Arm, Phase II Study to Assess Efficacy and Safety of Myrcludex B in Combination With Peginterferon Alfa-2a Versus Peginterferon Alfa-2a Alone in Patients With Chronic Viral Hepatitis B With Delta-agent
Brief Title: Myrcludex B in Combination With Peginterferon Alfa-2a Versus Peginterferon Alfa-2a Alone in Patients With Chronic Viral Hepatitis B With Delta-agent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hepatera Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYR 203
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-03

CONDITIONS: Chronic Viral Hepatitis B With Delta-agent
MeSH Terms: interventions — myrcludex-B; bulevirtide; peginterferon alfa-2a; Tenofovir

STUDY DESIGN:
Intervention Model Description: Multicenter, Open-label, Randomized, Comparative, parallel-arm phase II study
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm A (Active Comparator): PEG IFN alfa-2a 180 µg for 48 weeks
  Interventions: Drug: PEG IFN alfa-2a
- Arm B (Experimental): Myrcludex B 2 mg + PEG IFN alfa-2a 180 µg for 48 weeks
  Interventions: Drug: Myrcludex B; Drug: PEG IFN alfa-2a
- Arm C (Experimental): Myrcludex B 5 mg + PEG IFN alfa-2a 180 µg for 48 weeks
  Interventions: Drug: Myrcludex B; Drug: PEG IFN alfa-2a
- Arm D (Experimental): Myrcludex B 2 mg for 48 weeks
  Interventions: Drug: Myrcludex B
- Arm E (Experimental): Myrcludex B 10 mg (10 mg once a day) + PEG-IFN alfa-2a 180 μg during 48 weeks
  Interventions: Drug: Myrcludex B; Drug: PEG IFN alfa-2a
- Arm F (Experimental): Myrcludex B 10 mg (5 mg twice a day) + Tenofovir during 48 weeks
  Interventions: Drug: Myrcludex B; Drug: Tenofovir

INTERVENTIONS:
Drug: Myrcludex B — Lyophilised powder for solution for subcutaneous injection
  Other Names: Bulevirtide
  Arms: Arm B; Arm C; Arm D; Arm E; Arm F
Drug: PEG IFN alfa-2a — solution for subcutaneous injection, once per week
  Other Names: Pegasys
  Arms: Arm A; Arm B; Arm C; Arm E
Drug: Tenofovir — Film-coated tablets, 300 mg, per os, once daily
  Other Names: Viread
  Arms: Arm F

SUMMARY:
Randomised, Comparative, Parallel-Arm Study to Assess Efficacy and Safety of Myrcludex B in Combination with Peginterferon Alfa-2a Versus Peginterferon Alfa-2a Alone in Patients with Chronic Viral Hepatitis B with Delta-agent

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomised, comparative, active-controlled parallel-arm phase II study.

The study will be conducted in Russia. The aim of this study is to explore the safety and efficacy of treatment with Myrcludex B used as a monotherapy and in combination with PEG-IFNα and Tenofovir compared to monotherapy with PEG-IFNα in patients with chronic viral hepatitis B with delta-agent, based on the achievement of undetectable viral load at the end of the follow-up period 6 months (24 weeks) after the end of treatment. The study is also aimed at investigating immunogenicity of Myrcludex B and the drug pharmacokinetics when used in combination with PEG IFN alfa-2a and with Tenofovir.

It is planned to screen 110 patients, and 90 patients will be randomised in equal numbers into six treatment arms.

* Arm A (n=15): PEG IFN alfa-2a 180 µg for 48 weeks
* Arm B (n=15): Myrcludex B 2 mg + PEG IFN alfa-2a 180 µg for 48 weeks
* Arm C (n=15): Myrcludex B 5 mg + PEG IFN alfa-2a 180 µg for 48 weeks
* Arm D (n=15): Myrcludex B 2 mg for 48 weeks
* Arm E (n=15): Myrcludex B 10 mg (10 mg once a day)+ PEG IFN alfa-2a 180 µg for 48 weeks
* Arm F (n=15): Myrcludex B 10 mg (5 mg twice a day)+ Tenofovir for 48 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent form.
2. Males and females 18 to 65 years of age (inclusively).
3. Patients with chronic hepatitis B (HBeAg-positive or negative) and HBsAg-positive for at least 6 months prior to Screening.
4. Positive for anti-HDV antibodies for at least 6 months prior to Screening.
5. HDV RNA-positive at Screening.
6. ALT ≥ 1 x ULN and < 10 x ULN.
7. The patient agreed to use adequate method of contraception during the study, starting from the time of Informed Consent signing and until completion of the Follow-up Period.

Exclusion Criteria:

1. Intolerance or hypersensitivity to the active ingredient or other components of the study drug Myrcludex B.
2. Intolerance or hypersensitivity to interferons alfa, genetically engineered E.coli medications, polyethylene glycol or other components of peginterferon alfa-2a.
3. Previous treatment with Myrcludex B (patients with previous exposure to interferon are eligible).
4. Therapy with antiviral drugs for chronic viral hepatitis B with delta-agent over the previous 6 months.
5. Therapy with anti-tumour agents (including radiotherapy) or immunomodulatory medications (including systemic glucocorticoids) over the previous 6 months.
6. The following laboratory test results at Screening:

   1. Hemoglobin < 100 g/L
   2. Leucocytes < 3000/µL
   3. Neutrophils < 1500/µL
   4. Platelets < 90000/µL
   5. Serum creatinine >1.5 x ULN.
7. Total bilirubin > 34.2 µM/L. Patients with higher total bilirubin may be enrolled upon consultation with the study Medical Monitor, if there is clear evidence that the elevated bilirubin is caused by Gilbert's syndrome.
8. Current or previous decompensated liver disease, including coagulopathy, hyperbilirubinemia, hepatic encephalopathy, hypoalbuminaemia, ascites, and oesophageal varices haemorrhage; Child-Pugh score of B/C or ≥6 points.
9. HCV or HIV coinfection (patients with anti-HCV antibodies and no HCV RNA at Screening are eligible).
10. Hepatocellular carcinoma.
11. Signs of drug- or alcohol-induced liver disease or any other medical conditions associated with chronic liver disease (e.g. autoimmune hepatitis, hemochromatosis, thalassaemia, alcoholic hepatitis, toxic liver disease).
12. Contraindications for liver biopsy.
13. Concurrent malignancy (current diagnosed or suspected malignancy; risk of a previous malignancy recurrence).
14. Severe decompensated cardiovascular diseases, including unstable and poorly controlled conditions, over 6 months before Screening.
15. History of poorly controlled thyroid conditions or clinically significant signs of thyroid dysfunction at Screening.
16. Previous or current severe renal failure or significant renal dysfunction at Screening.
17. Previous or current chronic pulmonary disease with respiratory distortion at Screening.
18. Previous or current severe retinopathy, significant ophthalmology disorders associated with diabetes mellitus or hypertension.
19. Previous or current severe psychiatric disorders at Screening (e.g. severe depressions, suicidal attempts, severe neuroses or cognitive disorders).
20. Previous or current endocrine disorders (hypoglycaemia, hyperglycaemia, diabetes mellitus) that are not adequately controlled at Screening.
21. History of visceral organ transplantation.
22. Signs of drug and/or alcohol dependence (80 g of alcohol/day for men and 40 g of alcohol/day for women) within 1 year before Screening.
23. History of immune disorders (e.g. idiopathic thrombocytopenic purpura, lupus erythematosus, sclerodermia, severe psoriasis, rheumatoid arthritis).
24. Need for concomitant use of glucocorticoids or myelotoxic agents.
25. Participation in another clinical study within 30 days prior to enrollment into this study.
26. Pregnant or breast-feeding females.
27. Any other condition that, in the opinion of Investigator, precludes the patient from taking part in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Bogomolov, PhD, Principal Investigator — Moscow Regional Research and Clinical Institute (MONIKI)
Locations (7):
- Russia (7):
  - State Budgetary educational institution of higher professional education "South Ural State Medical University" Ministry of healthcare, Chelyabinsk
  - State Budgetary Institution of healthcare "Specialized Clinical Infectious Diseases Hospital" Ministry of Health, Krasnodar
  - Moscow Regional Research and Clinical Institute, Moscow
  - Federal Budget Institution of Science "Central Research Institute of Epidemiology" of The Federal Service on Customers' Rights Protection and Human Well-being Surveillance, Moscow
  - LLC "Clinic of Modern Medicine", Moscow
  - Medical Company "Gepatolog" LLC, Samara
  - State Budgetary Institution of healthcare 'Stavropol regional clinical hospital', Stavropol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lampertico P, Bogomolov PO, Chulanov V, Stepanova T, Morozov V, Allweiss L, Dandri M, Burhenne J, Blank A, Ciesek S, Elsner C, Dittmer U, An Q, Manuilov D, Da BL, Flaherty JF, Urban S, Wedemeyer H. Phase 2 Randomised Study of Bulevirtide as Monotherapy or Combined With Peg-IFNalpha-2a as Treatment for Chronic Hepatitis Delta. Liver Int. 2025 Feb;45(2):e70008. doi: 10.1111/liv.70008. PMID 39853842
- [Derived] Asselah T, Lampertico P, Aleman S, Bourliere M, Streinu-Cercel A, Bogomolov P, Morozov V, Stepanova T, Lazar S, Manuilov D, Mercier RC, Tseng S, Ye L, Flaherty JF, Osinusi A, Da BL, Chee GM, Lau AH, Brunetto MR, Wedemeyer H. Bulevirtide Monotherapy Is Safe and Well Tolerated in Chronic Hepatitis Delta: An Integrated Safety Analysis of Bulevirtide Clinical Trials at Week 48. Liver Int. 2025 Apr;45(4):e16174. doi: 10.1111/liv.16174. Epub 2024 Dec 8. PMID 39648559
- [Derived] Allweiss L, Volmari A, Suri V, Wallin JJ, Flaherty JF, Manuilov D, Downie B, Lutgehetmann M, Bockmann JH, Urban S, Wedemeyer H, Dandri M. Blocking viral entry with bulevirtide reduces the number of HDV-infected hepatocytes in human liver biopsies. J Hepatol. 2024 Jun;80(6):882-891. doi: 10.1016/j.jhep.2024.01.035. Epub 2024 Feb 8. PMID 38340811

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Started | 15 | 15 | 15 | 15 | 15 | 15
Completed | 10 | 13 | 15 | 13 | 14 | 14
Not Completed | 5 | 2 | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of consent | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 15 | 15 | 90
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (7.0) | 37.1 (5.5) | 36.9 (7.5) | 42.0 (9.6) | 36.2 (7.2) | 34.3 (7.2) | 36.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 8 | 4 | 3 | 4 | 33
  Male | 5 | 11 | 7 | 11 | 12 | 11 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 14 | 15 | 15 | 15 | 14 | 15 | 88
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 15 | 15 | 15 | 15 | 15 | 15 | 90
Height [Mean (Standard Deviation); unit: cm] | 168.9 (6.8) | 172.5 (9.4) | 171.4 (6.0) | 174.6 (8.6) | 174.1 (8.2) | 173.5 (6.8) | 172.5 (7.7)
Body Weight [Mean (Standard Deviation); unit: kg] | 68.02 (14.61) | 74.29 (14.44) | 72.37 (11.55) | 82.95 (16.38) | 72.67 (10.01) | 70.53 (9.08) | 73.47 (13.43)
Body Mass Idex [Mean (Standard Deviation); unit: kg/m²] | 23.77 (4.68) | 24.83 (3.46) | 24.69 (4.18) | 27.02 (3.91) | 24.03 (3.21) | 23.48 (3.31) | 24.64 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Negative HDV RNA by PCR
Description: Negativation of HDV RNA by PCR (undetectable HDV RNA) at Week 72 (end of follow-up period)
Time Frame: 72 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
Percentage of participants | 0 [0.0 to 21.8] | 53.3 [26.6 to 78.7] | 26.7 [7.8 to 55.1] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 33.3 [11.8 to 61.6]
Statistical Analysis 1: Comparison: Arm A vs Arm B; The proportions of negative HDV RNA response at week 72 in each of the MXB treatment groups were compared with the control group of PEG-IFNα by using Fisher's exact test and by presenting exact unconditional 95%-confidence intervals (CI) based on scores for the proportion differences; Test type: Superiority; p = 0.0022, Fisher Exact
Statistical Analysis 2: Comparison: Arm A vs Arm C; Test type: Superiority; p = 0.0996, Fisher Exact
Statistical Analysis 3: Comparison: Arm A vs Arm D; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Arm A vs Arm E; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 5: Comparison: Arm A vs Arm F; Test type: Superiority; p = 0.0421, Fisher Exact

2. Secondary Outcome: Percentage of Patients With Negative HDV RNA by PCR
Description: Percentage of patients with negative HDV RNA by PCR (undetectable HDV RNA) at Weeks 24 and 48
Time Frame: 24 and 48 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Week 24 | 6.7 [0.2 to 31.9] | 60.0 [32.3 to 83.7] | 60.0 [32.3 to 83.7] | 13.3 [1.7 to 40.5] | 66.7 [38.4 to 88.2] | 26.7 [7.8 to 55.1]
  Week 48 | 13.3 [1.7 to 40.5] | 80.0 [51.9 to 95.7] | 86.7 [59.5 to 98.3] | 13.3 [1.7 to 40.5] | 80 [51.9 to 95.7] | 46.7 [21.3 to 73.4]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Week 24; Test type: Superiority; p = 0.0052, Fisher Exact
Statistical Analysis 2: Comparison: Arm A vs Arm C; Week 24; Test type: Superiority; p = 0.0052, Fisher Exact
Statistical Analysis 3: Comparison: Arm A vs Arm D; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Arm A vs Arm E; Week 24; Test type: Superiority; p = 0.0017, Fisher Exact
Statistical Analysis 5: Comparison: Arm A vs Arm F; Week 24; Test type: Superiority; p = 0.3295, Fisher Exact
Statistical Analysis 6: Comparison: Arm A vs Arm B; Week 48; Test type: Superiority; p = 0.0007, Fisher Exact
Statistical Analysis 7: Comparison: Arm A vs Arm C; Week 48; Test type: Superiority; p = 0.0001, Fisher Exact
Statistical Analysis 8: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 9: Comparison: Arm A vs Arm E; Week 48; Test type: Superiority; p = 0.0007, Fisher Exact
Statistical Analysis 10: Comparison: Arm A vs Arm F; Week 48; Test type: Superiority; p = 0.1086, Fisher Exact

3. Secondary Outcome: Percentage of Patients With Normalized ALT
Description: Percentage of patients with normalized ALT at Weeks 24, 48 and 72. ALT normalisation was defined as having an ALT value within the normal range (≤31 U/L for females and ≤41 U/L for males)
Time Frame: 24, 48 and 72 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Week 24: number analyzed (Participants) | 15 | 15 | 15 | 14 | 15 | 15
  Week 24 | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 20.0 [4.3 to 48.1] | 64.3 [35.1 to 87.2] | 20.0 [4.3 to 48.1] | 60.0 [32.3 to 83.7]
  Week 48 | 26.7 [7.8 to 55.1] | 26.7 [7.8 to 55.1] | 46.7 [21.3 to 73.4] | 73.3 [44.9 to 92.2] | 26.7 [7.8 to 55.1] | 40.0 [16.3 to 67.7]
  Week 72: number analyzed (Participants) | 10 | 13 | 15 | 13 | 14 | 14
  Week 72 | 10.0 [0.3 to 44.5] | 53.8 [25.1 to 80.8] | 33.3 [11.8 to 61.6] | 23.1 [5.0 to 53.8] | 35.7 [12.08 to 64.9] | 35.7 [12.8 to 64.9]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Arm A vs Arm C; Week 24; Test type: Superiority; p = 0.2241, Fisher Exact
Statistical Analysis 3: Comparison: Arm A vs Arm D; Week 24; Test type: Superiority; p = 0.0002, Fisher Exact
Statistical Analysis 4: Comparison: Arm A vs Arm E; Week 24; Test type: Superiority; p = 0.2241, Fisher Exact
Statistical Analysis 5: Comparison: Arm A vs Arm F; Week 24; Test type: Superiority; p = 0.0007, Fisher Exact
Statistical Analysis 6: Comparison: Arm A vs Arm B; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 7: Comparison: Arm A vs Arm C; Week 48; Test type: Superiority; p = 0.4497, Fisher Exact
Statistical Analysis 8: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 0.0268, Fisher Exact
Statistical Analysis 9: Comparison: Arm A vs Arm E; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 10: Comparison: Arm A vs Arm F; Week 48; Test type: Superiority; p = 0.6999, Fisher Exact
Statistical Analysis 11: Comparison: Arm A; Week 72; Test type: Superiority; p = 0.0743, Fisher Exact
Statistical Analysis 12: Comparison: Arm A vs Arm C; Week 72; Test type: Superiority; p = 0.3449, t-test, 1 sided
Statistical Analysis 13: Comparison: Arm A vs Arm D; Week 72; Test type: Superiority; p = 0.6036, Fisher Exact
Statistical Analysis 14: Comparison: Arm A vs Arm E; Week 72; Test type: Superiority; p = 0.3408, Fisher Exact
Statistical Analysis 15: Comparison: Arm A vs Arm F; Week 72; Test type: Superiority; p = 0.3408, Fisher Exact

4. Secondary Outcome: Percentage of Patients With Combined Response
Description: Combined response is defined as negative HDV RNA and ALT normalization at Weeks 24, 48, and 72. The criteria for combined response were HDV RNA value below LLoD (where LLoD=10 IU/ml) and ALT within normal range (≤31 U/L for females and ≤41 U/L for males)
Time Frame: 24, 48 and 72 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Week 24 | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 20.0 [4.3 to 48.1] | 13.3 [1.7 to 40.5] | 13.3 [1.7 to 40.5] | 13.3 [1.7 to 40.5]
  Week 48 | 6.7 [0.2 to 31.9] | 20.0 [4.3 to 48.1] | 33.3 [11.8 to 61.6] | 13.3 [1.7 to 40.5] | 20.0 [4.3 to 48.1] | 13.3 [1.7 to 40.5]
  Week 72 | 0 [0.0 to 21.8] | 46.7 [21.3 to 73.4] | 13.3 [1.7 to 40.5] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Arm A vs Arm C; Week 24; Test type: Superiority; p = 0.2241, Fisher Exact
Statistical Analysis 3: Comparison: Arm A vs Arm D; Week 24; Test type: Superiority; p = 0.4828, Fisher Exact
Statistical Analysis 4: Comparison: Arm A vs Arm E; Week 24; Test type: Superiority; p = 0.4828, Fisher Exact
Statistical Analysis 5: Comparison: Arm A vs Arm F; Week 24; Test type: Superiority; p = 0.4828, Fisher Exact
Statistical Analysis 6: Comparison: Arm A vs Arm B; Week 48; Test type: Superiority; p = 0.5977, Fisher Exact
Statistical Analysis 7: Comparison: Arm A vs Arm C; Week 48; Test type: Superiority; p = 0.1686, Fisher Exact
Statistical Analysis 8: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 9: Comparison: Arm A vs Arm E; Week 48; Test type: Superiority; p = 0.5977, Fisher Exact
Statistical Analysis 10: Comparison: Arm A vs Arm F; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 11: Comparison: Arm A vs Arm B; Week 72; Test type: Superiority; p = 0.0063, Fisher Exact
Statistical Analysis 12: Comparison: Arm A vs Arm C; Week 72; Test type: Superiority; p = 0.4828, Fisher Exact
Statistical Analysis 13: Comparison: Arm A vs Arm D; Week 72; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 14: Comparison: Arm A vs Arm E; Week 72; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 15: Comparison: Arm A vs Arm F; Week 72; Test type: Superiority; p = 0.4828, Fisher Exact

5. Secondary Outcome: Percentage of Patients With HВsAg Response
Description: HВsAg response was defined as HBsAg negativation or > 1 log10 IU/mL decline from baseline.
Time Frame: 24, 48 and 72 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Week 24 | 6.7 [0.2 to 31.9] | 40.0 [16.3 to 67.7] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9]
  Week 48 | 0 [0.0 to 21.8] | 46.7 [21.3 to 73.4] | 20.0 [4.3 to 48.1] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8]
  Week 72 | 0 [0.0 to 21.8] | 40.0 [16.3 to 67.7] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Week 24; Test type: Superiority; p = 0.0801, Fisher Exact
Statistical Analysis 2: Comparison: Arm A vs Arm C; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Arm A vs Arm D; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Arm A vs Arm E; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 5: Comparison: Arm A vs Arm F; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 6: Comparison: Arm A vs Arm B; Week 48; Test type: Superiority; p = 0.0063, Fisher Exact
Statistical Analysis 7: Comparison: Arm A vs Arm C; Week 48; Test type: Superiority; p = 0.2241, Fisher Exact
Statistical Analysis 8: Comparison: Arm A vs Arm E; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 9: Comparison: Arm A vs Arm B; Week 72; Test type: Superiority; p = 0.0169, Regression, Cox
Statistical Analysis 10: Comparison: Arm A vs Arm C; Week 72; Test type: Superiority; p = 0.4828, Fisher Exact
Statistical Analysis 11: Comparison: Arm A vs Arm E; Week 72; Test type: Superiority; p = 0.4828, Fisher Exact

6. Secondary Outcome: Percentage of Patients With HBsAg Negativation
Description: Undetectable HВsAg with appearance of HbsAg antibodies or without it.
Time Frame: 48 and 72 weeks
Population: According to SAP Section 7.1.5 - Handling of missing data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Week 48 HBsAg negativation with appearance of HbsAg antibodies | 0 [0.0 to 21.8] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8]
  Week 72 HBsAg negativation with appearance of HbsAg antibodies: number analyzed (Participants) | 10 | 13 | 15 | 12 | 14 | 14
  Week 72 HBsAg negativation with appearance of HbsAg antibodies | 0 [0.0 to 30.8] | 23.1 [5.0 to 53.8] | 0 [0.0 to 21.8] | 0 [0.0 to 26.5] | 7.1 [0.2 to 33.9] | 0 [0.0 to 23.2]
  Week 48 HBsAg negativation without appearance of HbsAg antibodies | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Week 72 HBsAg negativation without appearance of HbsAg antibodies | 0 [0.0 to 30.8] | 7.7 [0.2 to 36.0] | 0 [0.0 to 21.8] | 0 [0.0 to 26.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Week 48; Test type: Superiority; p = 0.4828, Fisher Exact
Statistical Analysis 2: Comparison: Arm A vs Arm E; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Arm A vs Arm B; Week 72; Test type: Superiority; p = 0.2292, Fisher Exact
Statistical Analysis 4: Comparison: Arm A vs Arm E; Week 72; Test type: Superiority; p = 1.0000, Fisher Exact

7. Secondary Outcome: Percentage of Patients With Negative HBV DNA by PCR
Description: Percentage of patients with undetectable HBV DNA by PCR at Weeks 24, 48 and 72
Time Frame: 24, 48 and 72 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Week 24 | 33.3 [11.8 to 61.6] | 53.3 [26.6 to 78.7] | 40.0 [16.3 to 67.7] | 33.3 [11.8 to 61.6] | 53.3 [26.6 to 78.7] | 80.0 [51.9 to 95.7]
  Week 48 | 26.7 [7.8 to 55.1] | 73.3 [44.9 to 92.2] | 40.0 [16.3 to 67.7] | 33.3 [11.8 to 61.6] | 66.7 [38.4 to 88.2] | 93.3 [68.1 to 99.8]
  Week 72 | 33.3 [11.8 to 61.6] | 66.7 [38.4 to 88.2] | 40.0 [16.3 to 67.7] | 40.0 [16.3 to 67.7] | 26.7 [7.8 to 55.1] | 46.7 [21.3 to 73.4]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Week 24; Test type: Superiority; p = 0.4621, Fisher Exact
Statistical Analysis 2: Comparison: Arm A vs Arm C; Week 24; Test type: Superiority; p = 1.0000, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Arm A vs Arm D; Week 24; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Arm A vs Arm E; Week 24; Test type: Superiority; p = 0.4621, Fisher Exact
Statistical Analysis 5: Comparison: Arm A vs Arm F; Week 24; Test type: Superiority; p = 0.0253, Fisher Exact
Statistical Analysis 6: Comparison: Arm A vs Arm B; Week 48; Test type: Superiority; p = 0.0268, Fisher Exact
Statistical Analysis 7: Comparison: Arm A vs Arm C; Week 48; Test type: Superiority; p = 0.6999, Fisher Exact
Statistical Analysis 8: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 9: Comparison: Arm A vs Arm E; Week 48; Test type: Superiority; p = 0.0656, Fisher Exact
Statistical Analysis 10: Comparison: Arm A vs Arm F; Week 48; Test type: Superiority; p = 0.0005, Fisher Exact
Statistical Analysis 11: Comparison: Arm A vs Arm B; Week 72; Test type: Superiority; p = 0.1431, Fisher Exact
Statistical Analysis 12: Comparison: Arm A vs Arm C; Week 72; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 13: Comparison: Arm A vs Arm D; Week 72; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 14: Comparison: Arm A vs Arm E; Week 72; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 15: Comparison: Arm A vs Arm F; Week 72; Test type: Superiority; p = 0.7104, Fisher Exact

8. Secondary Outcome: The Intensity of Liver Fibrosis Based on Results of Transient Elastometry of Liver at Weeks 48 and 72.
Description: Change in liver stiffness and intensity of liver fibrosis based on results of transient elastometry of liver at weeks 48 and 72.
Time Frame: 48 and 72 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 13 | 13 | 14 | 9 | 15 | 15
kPa
  Change from baseline to Week 48 | -0.67 (2.78) | 1.97 (3.94) | -0.27 (3.83) | -0.66 (2.52) | -2.35 (7.47) | -1.12 (3.23)
  Change from baseline to Week 72: number analyzed (Participants) | 9 | 12 | 14 | 8 | 14 | 14
  Change from baseline to Week 72 | -0.67 (5.25) | 0.65 (2.10) | -2.06 (4.49) | 0.00 (6.19) | 0.21 (6.53) | -1.20 (2.68)

9. Secondary Outcome: Number of Participants With Change (Improvement / Worsening) in Fibrosis and Histological Activity Stage From Baseline to Post-treatment
Description: Change (improvement/ worsening) in fibrosis and histological activity stage according to the liver biopsy study results from baseline to post-treatment Liver fibrosis was evaluated by histological staging systems with stage 0 corresponding to absence of fibrosis and with the highest score (the last stage in all systems) corresponding to cirrhosis.
  Improvement is defined as a decrease of at least 1 point in histological staging systems; worsening is defined as an increase of at least 1 point.
  Data should be interpreted with caution due to low number of paired biopsies available.
Time Frame: 72 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 4 | 4 | 4 | 7 | 5 | 14
Participants
  Ishak fibrosis score: Improvement | 0 | 0 | 1 | 4 | 3 | 8
  Ishak fibrosis score: No change | 2 | 0 | 3 | 2 | 1 | 2
  Ishak fibrosis score: Worsening | 2 | 4 | 0 | 1 | 1 | 4
  Knodell fibrosis score: Improvement | 0 | 0 | 1 | 3 | 1 | 7
  Knodell fibrosis score: No change | 2 | 0 | 3 | 2 | 3 | 3
  Knodell fibrosis score: Worsening | 2 | 4 | 0 | 2 | 1 | 4
  Metavir fibrosis stage: Improvement | 0 | 0 | 1 | 4 | 1 | 7
  Metavir fibrosis stage: No change | 2 | 1 | 3 | 2 | 3 | 3
  Metavir fibrosis stage: Worsening | 2 | 3 | 0 | 1 | 1 | 4
  Metavir activity grade: Improvement | 1 | 1 | 2 | 6 | 1 | 8
  Metavir activity grade: No change | 2 | 1 | 2 | 1 | 3 | 5
  Metavir activity grade: Worsening | 1 | 2 | 0 | 0 | 1 | 1
  Histological activity index: Improvement | 2 | 1 | 2 | 6 | 2 | 9
  Histological activity index: No change | 0 | 0 | 2 | 1 | 1 | 1
  Histological activity index: Worsening | 2 | 3 | 0 | 0 | 2 | 4

10. Secondary Outcome: Change in Molecular Analyses of Relative HDV RNA Expression, Relative HBV Pregenomic Expression, Relative Total HBV RNA Expression (X Region), Relative HBV RNA Expression (S Region).
Description: Molecular analyses of relative HDV RNA expression, relative HBV pregenomic expression, relative total HBV RNA expression (X region), relative HBV RNA expression (S region) from baseline to post-treatment.
  *Biopsy post treatment performed at Week 48 for arm D:MXB 2mg and arm F:MXB 5mg bid + Tenofovir, and performed at Week 72 for arms A:PEG-IFN, B:MXB 2mg + PEG-IFN, C:MXB 5mg + PEG-IFN and arm E:MXB 10mg + PEG-IFN.
Time Frame: 48 and 72 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Relative value
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 4 | 4 | 3 | 6 | 5 | 14
Relative value
  Relative HDV RNA expression | -0.062 (0.097) | -0.068 (0.145) | 0.296 (0.652) | -1.220 (1.285) | -1.676 (2.754) | -0.975 (1.732)
  Relative HBV pregenomic expression | -0.028 (0.044) | -0.004 (0.007) | 0.003 (0.010) | -0.001 (0.006) | -0.041 (0.101) | 0.049 (0.257)
  Relative total HBV RNA expression (X region) | 0.080 (1.070) | -1.088 (1.624) | -1.295 (0.511) | -0.282 (0.796) | 0.160 (1.380) | 0.403 (1.477)
  Relative HBV RNA expression (S region) | -0.688 (1.977) | -2.295 (2.306) | -1.696 (1.423) | -0.451 (0.962) | 0.223 (1.909) | 0.733 (2.372)

11. Secondary Outcome: Change in Molecular Analyses of Total HBV DNA (X Region) Copies/Cell, HBV DNA (S Region) Copies/Cell, cccDNA Copies/Cell From Baseline to Post-treatment.
Description: Molecular analyses of total HBV DNA (X region) copies/cell, HBV DNA (S region) copies/cell, cccDNA copies/cell from baseline to post-treatment.
  *Biopsy post treatment performed at Week 48 for arm D:MXB 2mg and arm F:MXB 5mg bid + Tenofovir, and performed at Week 72 for arms A:PEG-IFN, B:MXB 2mg + PEG-IFN, C:MXB 5mg + PEG-IFN and arm E:MXB 10mg + PEG-IFN.
Time Frame: 48 and 72 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Copies/cell
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 4 | 4 | 3 | 6 | 5 | 14
Copies/cell
  Total HBV DNA (X region) copies/cell | -0.041 (0.215) | -0.027 (0.452) | -0.132 (0.223) | 0.036 (0.240) | -0.297 (0.874) | 0.087 (0.156)
  HBV DNA (S region) copies/cell | -0.413 (0.784) | -0.944 (1.265) | -0.747 (1.149) | 0.124 (0.954) | -1.545 (3.047) | 0.196 (0.517)
  cccDNA copies/cell | -0.045 (0.083) | 0.030 (0.050) | 0.004 (0.042) | -0.003 (0.200) | -0.117 (0.194) | 0.058 (0.165)

12. Secondary Outcome: Change in Molecular Analysis of HDAg Positive Hepatocytes (%) From Baseline to Post-treatment
Description: Molecular analysis of HDAg positive Hepatocytes (percentage of HDAg positive Hepatocytes) from baseline to post-treatment.
  *Biopsy post treatment performed at Week 48 for arm D:MXB 2mg and arm F:MXB 5mg bid + Tenofovir, and performed at Week 72 for arms A:PEG-IFN, B:MXB 2mg + PEG-IFN, C:MXB 5mg + PEG-IFN and arm E:MXB 10mg + PEG-IFN.
Time Frame: 48 and 72 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 4 | 3 | 2 | 5 | 5 | 14
Percentage
  Baseline | 0.757 (0.873) | 2.178 (3.275) | 1.209 (1.001) | 7.550 (7.905) | 12.521 (13.855) | 3.641 (5.919)
  Change from baseline to post-treatment: number analyzed (Participants) | 1 | 3 | 2 | 3 | 5 | 14
  Change from baseline to post-treatment | 0.099 (NA) — SD is not available as only one sample from the arm was anlyzed | -1.961 (3.439) | -1.134 (0.995) | -10.334 (9.041) | -9.028 (16.100) | -3.616 (5.923)

13. Secondary Outcome: Change in the Gene Expression Analyses From Baseline to Post-treatment
Description: Change in the gene expression analyses of CXCL10, NTCP, CYP7A1, ISG15, MX1, OAS, HLA-E, TAP1 and USP18 from baseline to post-treatment.
  Biopsy post treatment performed at Week 48 for arm D:MXB 2mg and arm F:MXB 5mg bid + Tenofovir, and performed at Week 72 for arms A:PEG-IFN, B:MXB 2mg + PEG-IFN, C:MXB 5mg + PEG-IFN and arm E:MXB 10mg + PEG-IFN.
Time Frame: Weeks 48 - 72
Population: FAS
Measure: Mean (Standard Deviation); unit: Relative value
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 5 | 14
Relative value
  CXCL10 relative expression | -0.017 (0.033) | -0.012 (0.019) | 0.010 (0.005) | -0.034 (0.009) | 0.003 (0.062) | -0.015 (0.017)
  NTCP relative expression | 0.001 (0.010) | -0.016 (0.012) | 0.001 (0.004) | 0.002 (0.005) | 0.011 (0.008) | 0.004 (0.008)
  CYP7A1 relative expression | 0.002 (0.006) | 0.002 (0.006) | 0.000 (0.001) | 0.001 (0.002) | -0.001 (0.002) | 0.001 (0.003)
  ISG15 relative expression | 0.207 (0.160) | -0.092 (0.321) | -0.003 (0.004) | -0.037 (0.024) | -0.163 (0.286) | -0.005 (0.034)
  MX1 relative expression | 0.175 (0.141) | -0.020 (0.186) | -0.013 (0.014) | -0.034 (0.019) | -0.056 (0.122) | -0.000 (0.026)
  OAS relative expression | 0.067 (0.059) | -0.019 (0.063) | 0.005 (0.009) | -0.015 (0.010) | -0.025 (0.049) | 0.003 (0.014)
  HLA-E relative expression | 0.038 (0.095) | -0.322 (0.175) | 0.015 (0.179) | -0.386 (0.197) | 0.149 (0.308) | -0.061 (0.191)
  TAP1 relative expression | 0.000 (0.007) | -0.012 (0.008) | -0.001 (0.004) | -0.017 (0.009) | 0.007 (0.019) | -0.004 (0.007)
  USP18 relative expression | 0.021 (0.017) | -0.003 (0.016) | -0.003 (0.006) | -0.005 (0.004) | -0.002 (0.012) | 0.001 (0.003)

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 13/15 | 14/15 | 14/15 | 15/15 | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=15) | Arm B (N=15) | Arm C (N=15) | Arm D (N=15) | Arm E (N=15) | Arm F (N=15)
Anal fistula (Gastrointestinal disorders) | NA | 1 (1) | NA | NA | NA | NA
Proctitis (Gastrointestinal disorders) | NA | 1 (1) | NA | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=15) | Arm B (N=15) | Arm C (N=15) | Arm D (N=15) | Arm E (N=15) | Arm F (N=15)
Total bile acids increased (Investigations) | 5 (18) | 10 (21) | 9 (31) | 12 (22) | 15 (45) | 15 (53)
ALT increased (Investigations) | 5 (11) | 5 (9) | 6 (11) | 8 (8) | 8 (24) | 4 (8)
AST increased (Investigations) | 5 (11) | 4 (8) | 4 (6) | 8 (8) | 6 (19) | 4 (5)
GGT increased (Investigations) | 4 (9) | 4 (7) | 3 (5) | 4 (5) | 8 (16) | 0 (0)
Haemoglobin decreased (Investigations) | 4 (5) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 2 (8) | 2 (4)
White blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (5) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (8) | 2 (4)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (2)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (2)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reticulocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time shortened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroxine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutripenia (Blood and lymphatic system disorders) | 8 (32) | 10 (28) | 9 (28) | 3 (6) | 14 (57) | 3 (12)
Leukopenia (Investigations) | 9 (25) | 8 (21) | 7 (19) | 4 (8) | 14 (58) | 4 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (16) | 11 (23) | 7 (18) | 3 (7) | 12 (29) | 5 (14)
Lymphopenia (Blood and lymphatic system disorders) | 5 (12) | 1 (1) | 1 (2) | 1 (1) | 5 (10) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 2 (4) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Reticulocytopenia (Blood and lymphatic system disorders) | 5 (12) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Erythropenia (Blood and lymphatic system disorders) | 4 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Reticulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (3) | 1 (2)
Monocytopenia (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic calcification (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 9 (11) | 8 (8) | 0 (0) | 3 (4) | 0 (0)
Asthenia (General disorders) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 1 (3)
Hyperthermia (General disorders) | 7 (26) | 0 (0) | 1 (5) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (8) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (6) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (5)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (8) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 2 (3)
Somnolence (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory track infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory track infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purulent discharge (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubineamia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 3 (7) | 2 (4)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic calcification (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fybromyalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02888106/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT02888106/SAP_001.pdf